CLINICAL TRIAL: NCT03103932
Title: BiomarkeR cAndidates to Guide Discharge of Patients Admitted to Hospital With heARt Failure
Brief Title: Biomarker Guided Discharge of Heart Failure Patients
Acronym: RADAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peter Liu (Other)
Collaborators: Genome Canada (Other); Roche Diagnostics GmbH (Industry); Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor-Investigator, Peter Liu, Chief Scientific Officer and VP of Research, Ottawa Heart Institute Research Corporation
Organization: Ottawa Heart Institute Research Corporation (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 806
Record Dates: First submitted 2017-03-28; First posted 2017-04-07 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Heart Failure; With Decompensation
Keywords: biomarkers; heart failure; hospital admission
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: single blind, strategy based, randomized trial consisting of two main study arms
Who Masked: Participant, Care Provider
Masking Description: The assigned care pathway will not be revealed to the participant NTproBNP levels will not be revealed to care providers for the group randomized to usual care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): Participants will be treated as is usual at each institution. Biomarkers will be measured on Day 2-3 and again prior to discharge from hospital. NTproBNP levels will not be revealed to care providers.
- Biomarker guided discharge pathway (Experimental): Admission NTproBNP levels will be used to stratify participants into lower and medium-higher risk care pathways. NTproBNP levels will be repeated on Day 2-3 and again prior to discharge. Each care pathway is designed to optimize discharge time according to NTproBNP levels. All NTproBNP results will be displayed on the front of the participant's chart along with the care pathway that the participant has been randomized to. The care providers will be reminded daily by the study team that the participant is in the biomarker guided discharge pathway arm of the study and that the designated care pathway should be followed as closely as possible.
  Interventions: Other: Biomarker guided discharge algorithm

INTERVENTIONS:
Other: Biomarker guided discharge algorithm — participants randomized to the biomarker guided discharge algorithm will follow a pre-determined care pathway for treatment of heart failure symptoms based on admission NTproBNP levels
  Arms: Biomarker guided discharge pathway

SUMMARY:
This is a multi-centre, single blind, randomized study. Patients admitted to hospital with acute decompensated heart failure will be randomized to biomarker guided discharge algorithm vs usual care in a 2:1 ratio. NTproBNP and other biomarkers will be measured within 24 hours of admission. The NTproBNP results will be used to further stratify participants randomized to the biomarker guided group into lower and medium to higher risk pathways. Biomarkers will be repeated after 2-3 days and again prior to discharge. Specific care pathways will be followed for each of the lower risk and medium-higher risk groups. Biomarkers will be repeated 30 days post discharge. Participants will be followed with a phone call at 3 months and return for a follow up visit at 6 months post discharge for outcome evaluation.

DETAILED DESCRIPTION:
Care Pathways:

Usual care: Participants will be treated for their heart failure symptoms as is usual at each participating institution. NTproBNP results will not be revealed to the care providers.

NTproBNP levels of participants randomized to the biomarker guided discharge algorithm will be posted on the participant's medical records. The results will be used by the care providers for decision making according to the predetermined care pathway.

Lower risk group: Participants who's admission NTproBNP is below 3,000 pg/ml will be placed into the lower risk group. Discharge planning will start within 24 hours of hospital admission. Symptoms will be treated aggressively. If the NTproBNP level drops to 1,500 pg/ml or below on Day 2-3, the participant will be discharged home. If the NTproBNP level does not drop to below 1,500 pg/ml, the participant will continue on treatment for another day or two and be discharged home when medically stabilized.

Medium-higher risk group: Participants who's admission NTproBNP is 3,000 pg/ml or above will be placed into the medium-higher risk group. Symptoms will be treated aggressively. If the NTproBNP level drops to below 3,000 pg/ml on Day 2-3, the participant will follow the lower risk pathway until discharge. If the NTproBNP level remains above 3,000 pg/ml, aggressive treatment of symptoms will continue. Biomarkers will be repeated on Day 6-7. If the NTproBNP level has dropped by at least 30% from admission and the participant is medically stabilized, the participant will be discharged home. If the NTproBNP level has not dropped by at least 30% from admission, treatment will continue until the participant is medically stabilized. This last group will be discharged home on telehealth with daily monitoring.

All participants will complete a Quality of Life questionnaire at admission and at the 30 day post discharge follow up.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to hospital with a primary diagnosis of acute decompensated heart failure, compatible with the modified Framingham criteria

Exclusion Criteria:

* Patient unable to provide blood samples or cannot participate in follow-up
* Patient with end stage organ failure

  * Kidney: creatinine >350 μmol/L or Estimated GFR ≤15 ml/min
  * Liver dysfunction: liver function test >2.5 times normal
  * Lungs: pulmonary FEV1<50% predicted
* Patient requiring intubation
* Patient with an admission NTproBNP measurement of >30,000 pg/ml
* Patient listed for heart transplant, or admitted specifically for transplant workup
* Patient in cardiogenic shock
* Patient with life expectancy of less than 6 months, or has major co-morbidities such as new stroke, cancer, pneumonia, or other serious life threatening illness
* Patient with conditions that will make it difficult to discharge from hospital such as a fall or waiting for a long term care bed
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the patient at risk because of participation in the trial, or may bias the result of the trial, or the patient's ability to participate in the trial
* Patient who has participated in another research trial involving an investigational product in the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2017-08-26 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
the total number of days alive and out of hospital during the first 30 days of heart failure diagnosis | Randomization to 30 days post randomization
  The investigator will measure te total number of days in hospital for each group
the total number of days alive and out of hospital during the first 30 days of heart failure diagnosis | Randomization to 30 days post randomization
  The investigator will measure the number of rehospitalizations in each group
the total number of days alive and out of hospital during the first 30 days of heart failure diagnosis | Randomization to 30 days post randomization
  The investigator will measure the total number of deaths and hospitalization episodes in each group

SECONDARY OUTCOMES:
the total number of days alive and out of hospital during the first 6 months of follow up | Randomization to 6 months post randomization
  The investigator will measure the total number of days in hospital in each group
the total number of days alive and out of hospital during the first 6 months of follow up | Randomization to 6 months post randomization
  The investigator will measure The number of rehospitalizations in each group
the total number of days alive and out of hospital during the first 6 months of follow up | Randomization to 6 months post randomization
  The investigator will measure the number of deaths/hospitalization episodes in each group

OTHER OUTCOMES:
Total cost savings for hospitalizations over the course of the study | From enrollment of first patient to completion of the study - expected to be about 2 years
  The investigator will measure the cost associated with each hospitalization in each group

CONTACTS AND LOCATIONS:
Overall Officials: Peter Liu, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
IPD will not be available to other researchers. Only results will be shared.